CLINICAL TRIAL: NCT01899833
Title: A Prospective, Open-label, Multicenter Study With Blinded Over-reading Characterizing the Efficacy and Safety of 99mTc-EC-DG in the Evaluation of Coronary Artery Disease (CAD)
Brief Title: Efficacy and Saftey Study of 99mTc-ECDG in the Evaluation of Coronary Artery Disease (CAD)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cell>Point LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-ECDG-C3
Record Dates: First submitted 2013-07-10; First posted 2013-07-16 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients receive typical imaging agent for rest and stress imaging then receive investigational imaging agent for rest and stress imaging
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 99mTc-EC-DG, Diagnostic (Experimental): 99mTc-EC-DG (25 ± 5 mCi, up to 250 µg EC-DG) will be administered by intravenous (IV) bolus injection. Other Name:Technetium-99m-labeled Ethylenedicysteine-Deoxyglucose
  Interventions: Diagnostic Test: 99mTc-Sestamibi

INTERVENTIONS:
Diagnostic Test: 99mTc-Sestamibi — An injection of 99mTC-Sestamibi will be administered by IV push under medically observed conditions.
  Other Names: 99mTc-Sestamibi (Mibi)

SUMMARY:
This study will compare how well a new radiolabeled imaging agent ECDG compares to the current testing for coronary artery disease (radiolabeled Sestamibi) during a rest and stress cardiac test as documented from results of a coronary angiogram (if performed).

DETAILED DESCRIPTION:
This study will be a prospective, open-label, multi-center study assessing the efficacy and safety of 99mTc-EC-DG compared to 99mTc-SPECT MPI imaging for detecting the presence, location, and severity of CAD as established by coronary angiography. Approximately 60 patients will be enrolled in the study.

Group 1 will be patients who have been evaluated for CAD within 3 to 30 days by any cardiovascular diagnostic imaging method (nuclear, ultrasound, CTA, MRI, etc.) and their physician has planned for coronary angiography but angiography has not yet been performed. In addition, the patient has not had coronary artery bypass graft (CABG). These patients can be enrolled.

Group 2 will be patients who have been evaluated for CAD within 3 to 30 days by any cardiovascular diagnostic imaging method (nuclear, ultrasound, CTA, MRI, etc.) and the patient has already had coronary angiography performed but has not received any coronary intervention subsequent to the procedure.

The following sequence of imaging procedures will be performed for both Group 1 and 2 patients: The first procedure will be a 99mTc-EC-DG rest study. This will be followed within 24 hours to 3 days with a 1-day protocol 99mTc-SPECT MPI rest/stress study. This will be followed within 24 hours to 3 days with a 99mTc-EC-DG stress study.

For both Group 1 and 2, if 1 of the diagnostic imaging procedures performed to evaluate the presence of CAD was a traditional 99mTc-SPECT MPI rest/stress study, this procedure must be repeated as 1 of the 3 SPECT imaging procedures required by the trial protocol.

The modality for provocative stress testing (exercise, pharmacologic, or exercise/pharmacologic) will be matched between the 99mTc-SPECT study and the 99mTc-EC-DG study. All prospectively performed 99mTc-EC-DG and 99mTc-SPECT studies will be conducted using regadenoson as the pharmacologic stress agent. All imaging studies (99mTc-EC-DG, 99mTc-SPECT, coronary angiography) will be over-read by blinded, trained reviewers. The consensus blinded read will determine and record the location of the CAD by relating the wall of the myocardium affected to include: anterior, Inferior, lateral, septal and apex. The angiography study will identify the arteries associated with the CAD; namely, left anterior descending, circumflex or right coronary arteries. The study will also determine the severity of the CAD by visually comparing the size and intensity of the ischemic signal on rest and stress images obtained approximately 15 and 60 minutes post injection.

The results from the consensus blinded read of coronary angiography will be considered truth for the presence, location, and severity of obstructive CAD and degree of stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Either of the following:

   1. Standard 99mTc-SPECT perfusion rest/stress study completed within 30 days prior to screening and a coronary angiography study is clinically planned after the 99mTc-C-DG rest and stress visits in this study
   2. Coronary angiography study planned or completed within 30 days of screening and no coronary intervention has been performed and willingness to complete a standard 99mTc-SPECT rest/stress study
3. The patient is able to provide informed consent to participate in this study
4. No change in medical therapy between study procedures.

Exclusion Criteria:

1. Known cardiomyopathy or history of congestive heart failure (CHF) due to left ventricular systolic dysfunction (ejection fraction < 40%)
2. Starting a new anti-anginal drug or performance of revascularization prior to completing the 99mTc-EC-DG rest and stress study visits
3. Contraindication for provocative stress testing based on American College of Cardiology/American Heart Association (ACC/AHA) guidelines for exercise or pharmacologic testing
4. Intolerance or inability to receive sestamibi, tetrofosmin, or regadenoson, or an inability or unwillingness to exercise on a graded treadmill or receive pharmacologic stress
5. Inability to lie still for approximately 30 minutes during image acquisition
6. Women of childbearing potential, unless willing to use adequate contraception throughout the duration of the trial. Adequate contraception is considered hormonal contraception for > 3 months prior to entry, intrauterine device (IUD) in place for at least 3 months, double barrier methods (condoms, diaphragm or spermicide), abstinence, or a partner with non-reversed vasectomy > 40 days prior to entry.
7. Pregnant or nursing
8. History of malignant disease (excluding treated basal cell or squamous cell carcinoma of skin, or low grade cancers that are stable and not interfering with exercise may be allowed with permission from the Medical Monitor) within 5 years prior to screening. Resolution of a prior malignancy more than 5 years prior to screening must be deemed as cured by the investigator
9. Any physical, psychological or substance abuse (drug or alcohol) condition which, in the opinion of the investigator, would interfere with the ability to provide informed consent or comply with study instructions or may adversely affect the safety of the patient if enrolled in this trial
10. A known allergy to 99mTc-EC-DG or its components
11. Inability to adhere to requirements specific to the study site's protocols for imaging and exercise/pharmacological stress testing, including but not limited to dietary restrictions and prohibited medications
12. Received an investigational drug within 30 days prior to this study
13. Prior bypass surgery
14. Enrolled or plans to enroll in another clinical trial during this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Characterization of the efficacy of 99mTCc-ECDG in the evaluation of Coronary Artery Disease | Visit 1a through Visit 3 approximately 3 to 20 days
  1. Determine efficacy (sensitivity and specificity) of 99mTc-ED-DG: i. Compare efficacy of a rest and stress study at approximately 15 minutes post injection compared with efficacy of a standard 99mTc-SPECT rest/stress perfusion study for detecting the presence of CAD using invasive coronary angiography as the truth standard.* ii. Compare efficacy of a rest and stress study at approximately 60 minutes post injection compared with a standard 99mTc-SPECT rest/stress perfusion study for detecting the presence of CAD using invasive coronary angiography as the truth standard.*
  * Images will be displayed using the standard Cedars Sinai tomographic display software which projects images in the short axis, vertical long, and horizontal long axis displays.

SECONDARY OUTCOMES:
Safety: The number of participants with Adverse Events | From screeniing through up to 14 days after last study related procedure
  Reported or observed Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Gary Heller, MD, Principal Investigator — Consultant
Locations (1):
- Tom Hennebry, MD, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No